CLINICAL TRIAL: NCT01958177
Title: Clinical Study to Evaluate the Safety and Efficacy of Bone Marrow Derived Mono Nuclear Stem Cell (BMMNCs) in Cerebellar Ataxia .It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Clinical Study to Evaluate the Safety and Efficacy BMMNC in Cerebellar Ataxia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, Co -investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC/BMCA/2013//01
Record Dates: First submitted 2013-07-31; First posted 2013-10-09 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Cerebellar Ataxia
Keywords: stem cell; cerebellar ataxia; BMMNC
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMMNC (Other): Intravenous transfer of of Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs)
  Interventions: Biological: Intravenous transfer of of Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs)

INTERVENTIONS:
Biological: Intravenous transfer of of Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs) — Total 3 doses ,in 30 days ,in 7days interval Intravenous transfer of of Bone Marrow derived Mono Nuclear Stem Cell BMMNCs)

SUMMARY:
Cerebellar ataxia is a complex motor disturbance, which, can occur as a result of many diseases and presents with symptoms of an inability to coordinate balance, gait, extremity and eye movements. Lesions to the cerebellum can cause dyssynergia, dysmetria, dysdiadochokinesia, dysarthria and ataxia of stance and gait. Deficits are observed with movements on the same side of the body as the lesion (ipsilaterally).

ELIGIBILITY:
Inclusion Criteria:

* Age limit: 18 -65
* Diagnosed as Cerebellar ataxia
* Willingness to undergo Bone marrow transplantation BMMNC.
* To give an informed consent as well as sign the required Informed Consent Form (ICF) for the study.
* willingness to regularly visit the hospital / clinic for follow up during the follow up period / on prior agreed time points as per the protocol.

Exclusion Criteria:

* Patients with pre-existing or current systemic disease such as lung , liver (exception: history of uncomplicated hepatitis A) gastrointestinal , cardiac, immunodeficiency (including HIV) or any other condition determined by history or laboratory investigation that could cause a neurological defect (including syphilis, clinically relevant polyneuropathy) etc.
* Women who are pregnant or lactating
* Chronic kidney disease due to autoimmune aetiology, connective tissue disease, amyloidosis and storage disorders.
* Suffering from Severe co-morbidities like cardiac insufficiency, congestive cardiac failure, malignancy, infection, sepsis and bed sores.
* Positive test results for HIV and AIDS complex ,HCV , HbsAg and Syphilis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
improve in INTERNATIONAL CO-OPERATIVE ATAXIA RATING SCALE | baseline and after 12 month
  To see improvement in INTERNATIONAL CO-OPERATIVE ATAXIA RATING SCALE when compare with baseline and after 12 month.

SECONDARY OUTCOMES:
Balance test | baseline and after 12 MONTH
  To see improvement in Balance test when compare with baseline and after 12 month.
Tremor Rating Scale | baseline and after 12 MONTH
  compare the pre and post Tremor Rating Scale
quality of life | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — Chaitanya Hospital
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India